CLINICAL TRIAL: NCT02265211
Title: Mindfulness and Acceptance-Based Treatments for Social Anxiety: Defusion App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilfrid Laurier University (Other)
Responsible Party: Principal Investigator, Meagan MacKenzie, Postdoctoral Fellow, Wilfrid Laurier University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4207
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Anxiety; Shyness
MeSH Terms: conditions — Anxiety Disorders; Shyness

ARMS (1):
- Self-Help App (Experimental): Smartphone app designed to teach cognitive defusion.
  Interventions: Behavioral: Self-Help App

INTERVENTIONS:
Behavioral: Self-Help App

SUMMARY:
This study evaluates a self-help app in the treatment of shyness and social anxiety in adults. All participants will be assigned to the treatment group. It is expected that using this app will result in a reduction in social anxiety.

DETAILED DESCRIPTION:
Over 2 million Canadians have suffered from social anxiety disorder (SAD) at some point in their lives. This disorder is characterized by a strong fear of negative evaluation in social situations and is associated with significant impairment in social interactions, educational/occupational achievement, and life satisfaction. Despite the fact that efficacious treatments have been developed and evaluated, both treatment effectiveness and treatment seeking behaviour remain below optimal levels. Combined with the many barriers to treatment (i.e., cost, stigma, access), researchers are investigating self-help modalities as an alternative to conventional psychotherapy.

The Defusion App is based on content from Fleming & Kocovski's (2013) self-help book "The Mindfulness & Acceptance Workbook for Social Anxiety & Shyness." Specifically, the app teaches users about the tendency of socially anxious individuals to fuse with their anxious thoughts (i.e., cognitive fusion), and strategies to reduce it.

In this experimental research study, a smartphone app designed to help with social anxiety and shyness will be evaluated for both effectiveness and frequency of use. The objectives will be to determine whether participants use the app, and whether use of the app is associated with a reduction in social anxiety.

Preliminary evidence has indicated that smartphone apps for mental health are associated with promising results. It is expected that the use of the app in the present research will be associated with reductions in social anxiety symptom severity and a greater use of cognitive defusion strategies.

The participants will be a community sample of individuals interested in seeking help with social anxiety and shyness as recruited by the use of posters around the Wilfrid Laurier University campus and in the community, as well as online.

ELIGIBILITY:
Inclusion Criteria:

* must be seeking help for shyness/social anxiety
* must own a smartphone

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Social Anxiety Interaction Scale at 7 days | Baseline and 7 days
  Self-reported social anxiety scores. Each item is scored 0 (not at all ) to 4 (extremely) yielding a total between 0 and 80.
Change from Baseline in Social Phobia Scale at 7 days | baseline and 7 days
  Self-reported social anxiety scores. Each item is scored 0 (not at all ) to 4 (extremely) yielding a total between 0 and 80.
Change from Baseline in Cognitive Fusion Questionnaire at 7 days | baseline and 7 days
  Self-reported cognitive fusion scores. Each item is scored 1 (never true ) to 7 (always true) yielding a total between 7 and 49.
Change from Baseline in Believability of Anxious Feelings and Thoughts Questionnaire at 7 days | baseline and 7 days
  Self-reported believability of anxious feelings and thoughts scores. Each item is scored 1 (not at all believable) to 7 (completely believable) yielding a total between 16 and 112.
Change from Baseline in Experiences Questionnaire at 7 days | baseline and 7 days
  Self-reported decentering scores. Each item is rated from 1 (never) to 5 (all the time) yielding a total between 20 and 100.
Change from Baseline in Brief Social Anxiety - Acceptance and Action Questionnaire at 7 days | baseline and 7 days
  Self-reported acceptance of social anxiety scores. Each item is rated from 1 (never true) to 5 (always true) yielding a total between 1 and 56..

SECONDARY OUTCOMES:
Readiness Ruler | baseline
  Self-reported readiness to change ruler. Participants indicate the degree to which they are ready to change on a visual analogue scale ranging from 0 (not prepared to change) to 10 (already changing).
Credibility/Expectancy Questionnaire | baseline
  Self-reported app credibility. Participants indicate how credible the treatment app seems.

CONTACTS AND LOCATIONS:
Overall Officials: Meagan B MacKenzie, Ph.D., Principal Investigator — Wilfrid Laurier University
Locations (1):
- Wilfrid Laurier University, Waterloo, Ontario, Canada